CLINICAL TRIAL: NCT04262323
Title: A Novel Mobile Phone Application for Blood Pressure Monitoring: A Comparison With the Oscillometric Brachial Cuff in Surgical Patients in the Postanesthesia Care Unit
Brief Title: A Novel Mobile Phone Application ( OptiBP) for Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Other Study IDs: P2020/081
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Technology
MeSH Terms: interventions — Blood Pressure Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: novel mobile phone application for blood pressure monitoring. — Comparative blood pressure measurement with the mobile phone application and the non-invasive reference method (upper arm cuff).

SUMMARY:
Evaluation of a novel mobile application designed to estimate blood pressure (systolic-diastolic and mean arterial pressure) based on collected optical signals on patient's finger treated in surgical patients in the post-anesthesia care unit

DETAILED DESCRIPTION:
The purpose of the study is to compare the blood pressure values measured by a novel mobile phone application ( camera of the smartphone will be obstructed by the patient's right index) and the values measured by reference method used (the oscillometric brachial cuff).

All patients scheduled for noncardiac surgery at Erasme Hospital Brussels, Belgium will be recruited and their pressure will be measured with both mesurement methods. (novel smartphone application versus upper arm cuff oscillometry) at 5 time points (each 20-30 minutes)

The OptiBP Application is a mobile application installed on a mobile phone which is a non-invasive data-logger intended to acquire physiological data from patients. By applying the patient's finger on a smartphone's camera, a movie is generated and transformed into values of diastolic, mean and systolic blood pressure.

Three measures will be taken (spaced by one minute) with both methods after a period of 3 minutes of rest at each time point.

The patient's blood pressure will be measured in parallel with the mobile application and with the reference equipment (the oscillometric brachial cuff).

Then, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the novel mobile application.

The goal is therefore to compare blood pressure values as obtained by the analysis of the data recorded by the OptiBP Mobile Application, against simultaneous measurements provided by the oscillometric brachial cuff

ELIGIBILITY:
Inclusion Criteria:

* Patients (Men or women) older than 18 years old scheduled for a noncardiac surgery and admiited in the post-anesthesia care unit after the surgery
* Informed Consent as documented by signature (signed before surgery)

Exclusion Criteria:

* Minor patients
* Patients unable to participate due to the illness.
* Patients that cannot sign informed consent
* Blood pressure difference between the two arms of more than10mmHg inter-arm difference)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the surgical department at Erasme hospital for a moderate risk surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Confirmation of Blood pressure values measured simultaneously with the novel mobile phone application | up to 2 hours
  Comparison of values to non-invasive reference method (the oscillometric brachial cuff )

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Study Chair — ERASME
Locations (1):
- Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Derived] Desebbe O, El Hilali M, Kouz K, Alexander B, Karam L, Chirnoaga D, Knebel JF, Degott J, Schoettker P, Michard F, Saugel B, Vincent JL, Joosten A. Evaluation of a new smartphone optical blood pressure application (OptiBP) in the post-anesthesia care unit: a method comparison study against the non-invasive automatic oscillometric brachial cuff as the reference method. J Clin Monit Comput. 2022 Oct;36(5):1525-1533. doi: 10.1007/s10877-021-00795-w. Epub 2022 Jan 3. PMID 34978654